CLINICAL TRIAL: NCT04262362
Title: The Frequency Of Sodium Hypochlorite Extrusion During Endodontic Treatments: A Clinical Study
Brief Title: The Frequency Of Sodium Hypochlorite Extrusion During Endodontic Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Mustafa Murat Koçak, Associate professor, Bulent Ecevit University
Other Study IDs: Bülent Ecevit universi
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Pain, Acute; Necrotic Pulp
MeSH Terms: conditions — Acute Pain; Dental Pulp Necrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Root canal treatment — Incidence of pain that may occur due to sodium hypochlorite extrusion

SUMMARY:
Sodium hypochlorite is a commonly used irrigation agent. However, the solution may extrude beyond the apex of tooth and cause pain during the treatment.The aim of this prospective observational investigation is to determinate the frequency of the extrusion of sodtium hypochlorite in endodontically treated teeth.

DETAILED DESCRIPTION:
Sodium hypochlorite (NaOCl) is a gold standard irrigation solution that has antimicrobial and tissue solvent effect. Until now, there is no other alternative that provides its activity characteristics. Although it represents many advantages, and it is usually considered safe, some cases of mishap and systematic reviews about case reports of NaOCl accident especially during endodontic procedures, have been reported in the literature. NaOCl may lead potentially very damaging injuring results with acute pain, swelling, hemolysis, ulceration, inhibition of neutrophil migration, endothelial and fibroblast cell damage, nerve weakness or damage, trismus and tissue necrosis if it overflows the periapical area.

The aim of this prospective observational investigation is to determinate the frequency of the extrusion in endodontically treated teeth.

The patients who applied to the clinic for dental treatment will be identified as having root canal treatment indication for at least one tooth. After the detailed medical and dental history will be obtained, the written consent form was taken from the patients who wanted to participate in the study. Age, gender, medical history, preoperative pain and pulpal status, having any periapical radiolusency of the related tooth will be recorded and root canal treatment will be performed according to routine procedures. After treatment, the code of tooth according to FDI classification, number of root, apical diameter, volume and concentration of irrigation solution will be recorded.

Routine treatment follow-up will be performed in patients who has no NaOCl overflow from the root during procedure. The patients with NaOCl overflow during the treatment process, appropriate treatment will be planned and followed up until symptoms regress.

ELIGIBILITY:
Inclusion Criteria:

* Requirement of root canal treatment

Exclusion Criteria:

* Sodium hypochlorite allergy
* Immature tooth
* root resorption

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient refer for routine endodontic treatment will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2020-09-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of pain and symptoms | During treatment
  pain or other symptoms due to sodium hypochlorite extrusion

CONTACTS AND LOCATIONS:
Locations (1):
- Bülent Ecevit University, Faculty of Dentistry, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No